CLINICAL TRIAL: NCT04909879
Title: Treatment of Non-COVID-19 Acute Respiratory Distress Syndrome: A Phase 2 Study of the Efficacy and Safety of Intravenous Allogeneic Adipose-Derived Mesenchymal Stem Cells
Brief Title: Study of Allogeneic Adipose-Derived Mesenchymal Stem Cells for Non-COVID-19 Acute Respiratory Distress Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Replaced by a different protocol.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-ARDS-201
Record Dates: First submitted 2021-05-29; First posted 2021-06-02 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Acute Respiratory Distress Syndrome; Ards
Keywords: ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-MSC (Experimental): Subjects will receive intravenous infusions of COVI-MSC (two vials or a total of ≈ 30 million cells) on Day 0, Day 2, and Day 4
  Interventions: Biological: COVI-MSC
- Placebo (Placebo Comparator): Subjects will receive intravenous infusions of placebo (two vials) on Day 0, Day 2, and Day 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-MSC — COVI-MSC are allogeneic culture-expanded adipose-derived mesenchymal stem cells
  Arms: COVI-MSC
Drug: Placebo — Excipient solution
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized study to assess the safety and efficacy of COVI-MSC in the setting of current standard of care treatments for subjects hospitalized subjects with acute respiratory distress syndrome not related to COVID-19 infection.

DETAILED DESCRIPTION:
This is a Phase 2, randomized controlled, multicenter study to assess the safety and efficacy of COVI-MSC in the setting of current standard of care treatments for subjects hospitalized subjects with acute respiratory distress syndrome not related to COVID-19 infection.

Subjects will be randomized 2:1 to receive COVI-MSC or placebo. COVI-MSC or placebo will be administered intravenously on Day 0, Day 2, and Day 4.

ELIGIBILITY:
Inclusion Criteria:

* Negative for SARS-CoV-2 infection as determined by an approved polymerase chain reaction (PCR) or an approved antigen test of any specimen
* Hospitalized with non-COVID-19-induced ARDS (any severity) with a PaO2/FiO2 (PF ratio) ≤ 300
* Requires oxygen supplementation at Screening
* Willing to follow contraception guidelines

Exclusion Criteria:

* Current standard of care treatments for ARDS appear to be working and the subject is clinically improving
* A previous stem cell infusion unrelated to this trial
* Pregnant or breast feeding or planning for either during the study
* Suspected uncontrolled active bacterial, fungal, viral, or other infection
* History of a splenectomy, lung transplant or lung lobectomy
* Concurrent participation in another clinical trial involving therapeutic interventions (observational study participation is acceptable)
* Expected survival or time to withdrawal of life-sustaining treatments expected to be < 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate at Day 28 | Baseline to Day 28
  All-cause mortality rate at Day 28

SECONDARY OUTCOMES:
All-cause mortality rate at Days 60 and 90 | Baseline to Day 60 and Day 90
  All-cause mortality rate at Days 60 and 90
Number of ventilator-free days through Day 28 | Baseline through Day 28
  Number of ventilator-free days through Day 28
Number of ICU days through Day 28 | Baseline through Day 28
  Number of ICU days through Day 28
Clinical status at Day 28 | Baseline to Day 28
  Clinical status as assessed using the Ordinal Scale for Clinical Improvement (0-8 scale, where lower score means better outcome)
Change in oxygenation | Baseline to Day 2, Day 4, Day 6, Day 14, Day 28
  Change in oxygenation at Days 2, 4, 6, 14, and 28 as measured using PaO2:FiO2 ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.